CLINICAL TRIAL: NCT00450398
Title: A Controlled, Prospective, Blinded, Randomized, Single-Center, Study of YSPSL for Prevention of Ischemic Reperfusion Injury in Patients Undergoing Cadaveric Orthotopic Liver Transplantation
Brief Title: YSPSL for Prevention of Delayed Graft Function in Cadaveric Liver Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Y's Therapeutics, Inc. (Industry)
Responsible Party: Stefan Hemmerich, PhD, RAC, Y's Therapeutics Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YSPSL-0002-PF
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Liver Diseases
Keywords: Delayed graft function
MeSH Terms: conditions — Liver Diseases; Delayed Graft Function | interventions — University of Wisconsin-lactobionate solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): YSPSL (rPSGL-Ig)
  Interventions: Drug: YSPSL
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YSPSL — YSPSL administered as an ex vivo flush (20 mg YSPSL in Viaspan® 200 mL total volume) into the portal vein prior to transplant at the back table; YSPSL 1 mg/kg administered IV to the transplant recipient prior to arterial reperfusion of the liver.
  Other Names: rPSGL-Ig; recombinant P-selectin glycoprotein ligand-Ig
  Arms: 1
Drug: Placebo — Ex vivo flush of placebo control (200 mL Viaspan®) into the portal vein prior to transplant and 0.1 mL/kg placebo control (saline) IV to the transplant recipient prior to arterial reperfusion of the liver.
  Other Names: Viaspan
  Arms: 2

SUMMARY:
The study is designed to assess the feasibility of evaluating YSPSL for the amelioration of ischemia reperfusion injury following liver transplantation by administering YSPSL into the liver graft directly ex vivo via the portal vein and to the recipient intravenously prior to reperfusion. Recently, P-selectin expression has been associated in liver grafts with prolonged cold storage times and rejection. By examining biomarkers of IRI including P-selectin by immunohistochemistry and/or quantitative PCR, liver histology and hepatic blood flow using established techniques, the goal of this study is to evaluate the feasibility of using these modalities for future studies of safety and efficacy.

DETAILED DESCRIPTION:
This will be a single-center, single-dose study. The study will be a randomized, double-blind, placebo-controlled, single-dose study. Patients who are undergoing cadaveric orthotopic liver transplantation and are at risk for development of DGF, based upon known risk factors, will be eligible to participate in the study. 12 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient will be a recipient of a primary (first) ABO compatible cadaveric liver allograft;
2. Patient's age is >=18 years;
3. Patient is not a recipient of a multivisceral transplant or simultaneous kidney transplant;
4. Patient has not undergone prior organ or cellular transplant of any type;
5. Patient has a Model for End Stage Liver Disease (MELD) score of <28;
6. Cold ischemia time (CIT) anticipated to be less than 12 hours;
7. Donor liver procured by UCLA liver team;
8. Veno-veno bypass is not planned to be used for the patient (e.g. no prior surgery or other factor that indicates a risk for excessive blood loss and therefore a need for veno-veno bypass +/- autologous recovery during surgery);
9. For patients who are women of childbearing potential, patient has a negative pregnancy test (either urine or serum) within 48 hours prior to transplant;
10. Patient (male and female) is willing to use an acceptable form of birth control for at least 3 months post-treatment; and
11. Patient is willing and able to sign informed consent.

Exclusion Criteria:

1. Patient has a prior organ transplant of any type;
2. Patient has known allergic or intolerance reactions to human immune globulins, antibodies, or components of the formulation or known contraindication to administration of YSPSL;
3. Patient has an uncontrolled active infection (on antibiotics with controlled infection is not an exclusion) ;
4. Patient has active Hepatitis B virus (HBV)/transplant for HBV related cirrhosis;
5. Patient has previously participated in this study or another study with YSPSL;
6. Patient has received investigational therapy within 90 days prior to the transplant procedure;
7. Patient has current drug or alcohol abuse or, in the opinion of the investigator, is at risk for poor compliance with the visits in this protocol (no drug testing required);
8. Patient is a pregnant or nursing female, a female of childbearing potential planning to become pregnant within the duration of this study, or is not practicing birth control;
9. Patient is planned to receive a living donor liver transplant;
10. Patient lives >200 miles away or otherwise is not able to participate in study follow-up visits;
11. Donor body mass index >28;
12. Donor liver biopsy >20% macrosteototic fat;
13. Donor age >65.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Delayed graft function post transplant | 6 months

SECONDARY OUTCOMES:
Liver function parameters through 6 months post transplant | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hemmerich, PhD, Study Director — Y's Therapeutics, Inc.
Locations (1):
- UCLA School of Medicine, Los Angeles, California, United States